CLINICAL TRIAL: NCT04677361
Title: A Pilot Study to Assess the Feasibility of Expanding Marrow Infiltrating Lymphocytes (MILs™) From Bone Marrow in Non-Small Cell Lung Cancer (NSCLC) and Small Cell Lung Cancer (SCLC) and Subsequently the Efficacy and Safety of MILs™ in Combination With Pembrolizumab in Patients With NSCLC and SCLC
Brief Title: Feasibility Study on Expandion of MILs From NSCLC and SCLC Patients and Infusion With Pembrolizumab
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Grantor shifted focus in disease, funding was stopped
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: WindMIL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-161; 20-1031 (Other: Fox Chase cancer Center)
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: SCLC; NSCLC
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Prior to treatment of MILs™ patients will receive non-myeloablative lymphodepletion with cyclophosphamide and fludarabine to increase the efficacy of adoptive T cell therapy. Bone marrow aspirate (BMA) will be collected from the patient to manufacture the MILs™. Upon progression and after the bone marrow is collected, a subject may receive bridging treatment of pembrolizumab until the MILs™ are received, after which treatment of the MILs™ and pembrolizumab will begin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MILs™ in Combination with Pembrolizumab (Experimental): Each patient will have their bone marrow collected, MILs produced, and the patient will be dosed with all of the MILs produced for that individual patient. The minimum requirement for treatment is 2 x 108 cells. The MILs™ must be administered via a central catheter which could either be a PICC line, port or central line.
  Subjects will be treated with MILs™ and pembrolizumab (200 mg Q3W) combination. MILs™ will be administered on Day 0 and pembrolizumab administered on Day 1. Pembrolizumab will be administered as a 30 minute IV infusion with a window of -5 minutes and +10 minutes is permitted.
  Interventions: Combination Product: MILs™ in Combination with Pembrolizumab

INTERVENTIONS:
Combination Product: MILs™ in Combination with Pembrolizumab — Efficacy and Safety of MILs™ in Combination with Pembrolizumab in Patients with NSCLC and SCLC

SUMMARY:
Marrow infiltrating lymphocytes (MILs™) are a novel method of adoptive cell therapy that provide an activated, polyclonal population of autologous tumor-specific T cells derived from the bone marrow. MILs™ in this study will be used to treat small cell lung cancer (SCLC) that has become resistant to chemotherapy and radiation.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is generally treated with surgery or chemotherapy, with or without radiation therapy, depending on staging. The problem with current available treatments is that SCLC almost always becomes resistant to chemotherapy and radiation. Marrow infiltrating lymphocytes (MILs™) are a novel method of adoptive cell therapy that provide an activated, polyclonal population of autologous tumor-specific T cells derived from bone marrow. Prior to treatment of MILs™ patients will receive non-myeloablative lymphodepletion with cyclophosphamide and fludarabine to increase the efficacy of adoptive T cell therapy. Bone marrow aspirate (BMA) will be collected from the patient to manufacture the MILs™. Upon progression and after the bone marrow is collected, a subject may receive bridging treatment of pembrolizumab until the MILs™ are received, after which treatment of the MILs™ and pembrolizumab will begin.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Patients must have histologically or cytologically confirmed SCLC or NSCLC.
3. Patients who have undergone chemotherapy must have had last dose ≥21 days prior to BMA; subjects who are currently being treated, bone marrow may be collected between cycles (prior to Day 1 of the next cycle).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 prior to BMA collection.
5. Willingness to complete a BMA.
6. Patients must have adequate bone marrow function prior to BMA collection:

   * Platelet count ≥ 100 × 109/L
   * Absolute neutrophil count (ANC) ≥ 1.0 ×109/L
   * Lymphocyte count ≥ 0.5 ×109/L
7. Patients must not have any history of coagulopathy or prothrombin time (PT)/partial thromboplastin time (PTT) > 2x upper limit of normal (ULN)(unless on an anticoagulant). If the patient is on an anticoagulant, it should be halted for 5 days prior to the BMA and PT/PTT < 2x ULN by the day of the procedure.
8. Ability to understand and willingness to sign a written informed consent and HIPAA consent document.

Exclusion Criteria:

1. Prior hematopoietic stem cell transplantation.
2. History of another primary malignancy that has been diagnosed or required therapy within the past 2 years prior to BMA collection (except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast).
3. Infection requiring treatment with antibiotics, antifungal, or antiviral agents within 7 days before the BMA.
4. Presence of an autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosis) requiring active systemic treatment. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are not excluded.
5. Clinically significant, uncontrolled cardiovascular disease, including congestive heart failure Grade III or IV according to the New York Heart Association classification, myocardial infarction, or unstable angina within the previous 6 months prior to BMA collection.
6. Major surgical procedure within 7 days of BMA. Procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures.
7. Administration of neutrophil growth factor support within 14 days prior to the BMA.
8. Prior radiation to both sides of the pelvis. Prior radiation to one side of the pelvis is permitted as long as the other side has not received radiation and is solely use to collect the bone marrow aspiration.
9. Use of systemic corticosteroids (glucocorticoids) for greater than one day within 28 days prior to the BMA. However, if a patient has an IV contrast allergy for CT, steroids should be used according to the institutional guidelines for contrast dye allergy.
10. Known diagnosis of human immunodeficiency virus (HIV) or active viral hepatitis, testing is not required.
11. Breast feeding females or pregnant females as documented by a serum beta human chorionic gonadotropin (β-hCG) pregnancy test consistent with pregnancy, obtained within 72 hours of BMA. Refer to section 5.4 for further detail.
12. Unwilling or unable to comply with the protocol (e.g., scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions)
13. Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of infusion of MILs™ by Adverse Events per | 2 years
  To assess the safety and tolerability of MILs™ in patients with NSCLC and SCLC

SECONDARY OUTCOMES:
Progression free survival (PFS) in patients as the length of time from the day of MILs™ administration to progression of the disease | 2 years
  To determine the efficacy per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 of MILs™ + pembrolizumab administration in patients with NSCLC and SCLC
Overall response rate (ORR) as the portion of patients with a tumor size reduction from the time of MILs™ administration to the time first response is seen in patients, whether it is partial response (PR) or complete response (CR | 2 years
  To determine the efficacy per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 of MILs™ + pembrolizumab administration in patients with NSCLC and SCLC

IPD SHARING:
Plan to Share IPD: No